CLINICAL TRIAL: NCT00887666
Title: Pilot Study: Hypovitaminosis D, Hyperparathyroidism and Hypomagnesemia in Patients With Congestive Heart Failure
Status: Completed | Type: Observational
Sponsor: State University of New York - Downstate Medical Center (Other)
Responsible Party: Mariana Markell, MD, SUNY Downstate Medical Center
Other Study IDs: 07-121
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Congestive Heart Failure; Hypovitaminosis D; Hyperparathyroidism
MeSH Terms: conditions — Heart Failure; Vitamin D Deficiency; Hyperparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
People with heart failure may have low magnesium and low vitamin D levels. They may also have abnormally high levels of parathyroid hormones. Magnesium and vitamin D are important chemicals that are not routinely measured in blood tests. We are studying how many people with heart failure have low levels of magnesium and vitamin D. We are also studying how many people with heart failure have overactive parathyroid glands and if that is related to their vitamin D levels.

DETAILED DESCRIPTION:
This is a single-encounter crossectional prevalence study in which demographic information, health opinion surveys and labwork are all obtained at one visit. There are no follow up visits, however, if abnormal lab results are discovered, participants will be notified via US mail.

ELIGIBILITY:
Inclusion Criteria:

* congestive heart failure

Exclusion Criteria:

* pregnant
* hospitalized within one month
* taking calcium, vitamin D or magnesium supplements
* proteinuria > 1g/24h
* creatinine clearance <35 (MDRD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with congestive heart failure
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of hypovitaminosis D, Hyperparathyroidism, Hypomagnesemia in our cohort of CHF patients | One year

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Markell, MD, Principal Investigator — State University of New York - Downstate Medical Center
Locations (1):
- SUNY Downstate Medical Center, Brooklyn, New York, United States